CLINICAL TRIAL: NCT04116333
Title: Effect of Using Endotracheal Tube Introducer for Intubation During Mechanical Chest Compressions in a Manikin: Randomized, Prospective, Crossover Study
Brief Title: Effect of Using Endotracheal Tube Introducer for Intubation During Mechanical Chest Compressions in a Manikin
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Derince Training and Research Hospital (Other)
Responsible Party: Principal Investigator, ASIM ENES ÖZBEK, Principal Investigator, Derince Training and Research Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2019-79
Record Dates: First submitted 2019-09-25; First posted 2019-10-04 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Intubation, Intratracheal; Advanced Cardiac Life Support

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to perform either Macintosh laryngoscope or Macintosh laryngoscope with endotracheal tube introducer first, using the envelope method. After completing these initial interventions, they will use the second method.
Who Masked: Participant
Masking Description: Participants will be aware of the general nature of the study, but they will be blinded to specific objectives of the study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ML + ETI (Experimental): Intubation with using endotracheal tube introducer with the Macintosh laryngoscope on a manikin during continuous chest compressions with mechanical compression device.
  Interventions: Device: Endotracheal tube introducer; Device: Macintosh laryngoscope
- ML (Active Comparator): Intubation with using the Macintosh laryngoscope on a manikin during continuous chest compressions with mechanical compression device.
  Interventions: Device: Macintosh laryngoscope

INTERVENTIONS:
Device: Endotracheal tube introducer — Use of endotracheal tube introducer with the Macintosh laryngoscope on a manikin during continuous chest compressions with mechanical compression device.
  Arms: ML + ETI
Device: Macintosh laryngoscope — Use of the Macintosh laryngoscope on a manikin during continuous chest compressions with mechanical compression device.

SUMMARY:
The aim of this study was to compare the impact of using ETI with the Macintosh laryngoscope on first pass success rates of the final year students of medical school on a manikin during continuous chest compressions with mechanical compression device.

DETAILED DESCRIPTION:
Fifty-two final year students of Kocaeli University Medical School will participate to the study. The participants will complete the one-hour training lecture on the use of the Macintosh laryngoscope (ML) and the endotracheal tube introducer (ETI) that will be instructed by an emergency medicine specialist. The information section will be followed by a chance of practice each endotracheal intubation method once by using the ML with and without the ETI on the manikin.

Mechanical compression device will be used to perform chest compressions. The manikin will be placed on an ambulance stretcher in a supine position. Airway interventions will be performed in a sitting position on a seat that will be adjusted to the same height with the ambulance seat. The airway kit will be placed beside the head of the manikin.

Each participant will perform 2 airway interventions. Participants will be allowed for maximum 2 attempts for each method. Each procedure will be recorded to the video camera. The participants will be aware of the video camera. Following the interventions each participant will be asked to grade the difficulty of the both methods on a 5-point Likert scale defined as 1: very easy, 2: easy, 3: moderate, 4: difficult and 5: very difficult. The participants will be asked for whether they have prior clinical experience or not with ML or/and ML with ETI use.

ELIGIBILITY:
Inclusion Criteria:

* Participants who want to participate the study

Exclusion Criteria:

* Participants who do not want to participate the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2019-10-09 (Estimated); Primary Completion 2019-10-10 (Estimated); Study Completion 2019-10-10 (Estimated)

PRIMARY OUTCOMES:
First pass success | 1 minute
  Comparison of the first pass success of the Macintosh laryngoscope and Macintosh laryngoscope with endotracheal tube introducer groups

SECONDARY OUTCOMES:
Time to endotracheal intubation | 1 minute
  The mean time to successful endotracheal intubation of Macintosh laryngoscope and Macintosh laryngoscope with endotracheal tube introducer groups
Second endotracheal intubation attempt success rates | 1 minute
  Second endotracheal intubation attempt success rates of Macintosh laryngoscope and Macintosh laryngoscope with endotracheal tube introducer groups
Difficulty level of each method according to the Likert scale | 1 minute
  Grading the difficulty of the Macintosh laryngoscope and Macintosh laryngoscope with endotracheal tube introducer on a 5-point Likert scale

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Benjamin EJ, Blaha MJ, Chiuve SE, Cushman M, Das SR, Deo R, de Ferranti SD, Floyd J, Fornage M, Gillespie C, Isasi CR, Jimenez MC, Jordan LC, Judd SE, Lackland D, Lichtman JH, Lisabeth L, Liu S, Longenecker CT, Mackey RH, Matsushita K, Mozaffarian D, Mussolino ME, Nasir K, Neumar RW, Palaniappan L, Pandey DK, Thiagarajan RR, Reeves MJ, Ritchey M, Rodriguez CJ, Roth GA, Rosamond WD, Sasson C, Towfighi A, Tsao CW, Turner MB, Virani SS, Voeks JH, Willey JZ, Wilkins JT, Wu JH, Alger HM, Wong SS, Muntner P; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2017 Update: A Report From the American Heart Association. Circulation. 2017 Mar 7;135(10):e146-e603. doi: 10.1161/CIR.0000000000000485. Epub 2017 Jan 25. No abstract available. Erratum In: Circulation. 2017 Mar 7;135(10):e646. doi: 10.1161/CIR.0000000000000491. Circulation. 2017 Sep 5;136(10):e196. doi: 10.1161/CIR.0000000000000530. PMID 28122885
- [Background] McNally B, Robb R, Mehta M, Vellano K, Valderrama AL, Yoon PW, Sasson C, Crouch A, Perez AB, Merritt R, Kellermann A; Centers for Disease Control and Prevention. Out-of-hospital cardiac arrest surveillance --- Cardiac Arrest Registry to Enhance Survival (CARES), United States, October 1, 2005--December 31, 2010. MMWR Surveill Summ. 2011 Jul 29;60(8):1-19. PMID 21796098
- [Background] Link MS, Berkow LC, Kudenchuk PJ, Halperin HR, Hess EP, Moitra VK, Neumar RW, O'Neil BJ, Paxton JH, Silvers SM, White RD, Yannopoulos D, Donnino MW. Part 7: Adult Advanced Cardiovascular Life Support: 2015 American Heart Association Guidelines Update for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2015 Nov 3;132(18 Suppl 2):S444-64. doi: 10.1161/CIR.0000000000000261. No abstract available. PMID 26472995
- [Background] Kleinman ME, Perkins GD, Bhanji F, Billi JE, Bray JE, Callaway CW, de Caen A, Finn JC, Hazinski MF, Lim SH, Maconochie I, Nadkarni V, Neumar RW, Nikolaou N, Nolan JP, Reis A, Sierra AF, Singletary EM, Soar J, Stanton D, Travers A, Welsford M, Zideman D. ILCOR Scientific Knowledge Gaps and Clinical Research Priorities for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care: A Consensus Statement. Circulation. 2018 May 29;137(22):e802-e819. doi: 10.1161/CIR.0000000000000561. Epub 2018 Apr 26. PMID 29700123
- [Background] Brooks SC, Anderson ML, Bruder E, Daya MR, Gaffney A, Otto CW, Singer AJ, Thiagarajan RR, Travers AH. Part 6: Alternative Techniques and Ancillary Devices for Cardiopulmonary Resuscitation: 2015 American Heart Association Guidelines Update for Cardiopulmonary Resuscitation and Emergency Cardiovascular Care. Circulation. 2015 Nov 3;132(18 Suppl 2):S436-43. doi: 10.1161/CIR.0000000000000260. No abstract available. PMID 26472994
- [Background] Le DH, Reed DB, Weinstein G, Gregory M, Brown LH. Paramedic use of endotracheal tube introducers for the difficult airway. Prehosp Emerg Care. 2001 Apr-Jun;5(2):155-8. doi: 10.1080/10903120190940038. PMID 11339725
- [Background] Kovacs G, Law JA, McCrossin C, Vu M, Leblanc D, Gao J. A comparison of a fiberoptic stylet and a bougie as adjuncts to direct laryngoscopy in a manikin-simulated difficult airway. Ann Emerg Med. 2007 Dec;50(6):676-85. doi: 10.1016/j.annemergmed.2007.05.022. Epub 2007 Aug 3. PMID 17681639
- [Background] Park L, Zeng I, Brainard A. Systematic review and meta-analysis of first-pass success rates in emergency department intubation: Creating a benchmark for emergency airway care. Emerg Med Australas. 2017 Feb;29(1):40-47. doi: 10.1111/1742-6723.12704. Epub 2016 Oct 27. PMID 27785883